CLINICAL TRIAL: NCT05844735
Title: A Two-part, Randomized Partially-blinded, Parallelgroup, Placebo- and Active Comparatorcontrolled Phase 1 Study to Evaluate the Photosafety of Repeated Oral Dose of SAR441566 in Healthy Adult Participants
Brief Title: A Randomized Placebo- and Active Comparator-controlled Study to Evaluate the Photosafety of SAR441566
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDY16917; U1111-1255-5054 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Applicable for Part I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part I SAR441566 Dose A (Experimental): Participants will receive repeated low dose of SAR441566 for 7.5 days
  Interventions: Drug: SAR441566
- Part I SAR441566 Dose B (Experimental): Participants will receive repeated high dose of SAR441566 for 7.5 days
  Interventions: Drug: SAR441566
- Part I Placebo (Placebo Comparator): Participants will receive repeated SAR441566 matching placebo tablets for 7.5 days
  Interventions: Drug: Placebo
- Part II Ciprofloxacin (Active Comparator): Participants will receive repeated ciprofloxacin 500 mg twice-daily (BID) for 5.5 days
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: SAR441566 — Tablet
  Arms: Part I SAR441566 Dose A; Part I SAR441566 Dose B
Drug: Placebo — Tablet
  Arms: Part I Placebo
Drug: Ciprofloxacin — Tablet
  Arms: Part II Ciprofloxacin

SUMMARY:
This is a single center randomized parallel-group partially-blinded, 4-arm Phase 1 study to evaluate the phototoxic potential of two dose levels of SAR441566 treatment compared to placebo and the active comparator, ciprofloxacin, in healthy adults, 18 to 55 years of age.

There will be two parts:

* Part I is a randomized placebo-controlled trial comparing sensitivity to ultraviolet (UV) light in participants treated with SAR441566 to those treated with placebo.
* Part II is an open label arm consisting of participants treated with ciprofloxacin which induces mild phototoxicity and serves as a positive control.

DETAILED DESCRIPTION:
The overall duration of the study for each participant will be up to approximately 48 days

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are between 18 and 55 years of age, (inclusive), at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* Participants with Fitzpatrick skin type classification of I, II, or III (I always burns easily, never tans, II always burns easily, tans minimally, III Burns moderately, tans gradually)
* Body weight within 50.0 and 100.0 kg (inclusive), and body mass index (BMI) within the range 18.0 and 32.0 kg/m2 (inclusive)

Exclusion Criteria:

* A positive hepatitis B (HBsAg, anti-HBc), hepatitis C or HIV test at screening, indicative of a current or past infection
* A history of active tuberculosis (TB) or positive serological test for TB (Quantiferon TB Gold or T-SPOT)
* History of invasive opportunistic infections
* Participants with a history of Clostridium difficile-associated diarrhea
* Participants with a history of malignancy occurring within 5 years before inclusion (except adequately treated carcinoma in situ of the cervix, or adequately treated non-metastatic squamous cell or basal cell carcinoma of the skin)
* Active skin disorders or alterations such as tattoos on the back where photosensitivity testing will be performed or unprotected ultraviolet exposure of the test areas within 4 weeks prior to baseline photo testing that the Investigator considers will interfere with study assessments
* Abnormal skin response during preliminary or baseline phototoxicity evaluations
* Any medication within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication (whichever is longer); any acetaminophen intake within 2 days prior the inclusion and any biologics (antibody or its derivatives) given within 4 months before screening
* Any participant enrolled or having participated, in this or any other clinical study involving an IMP or in any other type of medical research within the past 14 days (last day of IMP dosing in the previous clinical trial) or 5 half-lives whichever is longer, before screening
* Clinical signs and symptoms consistent with COVID-19 or laboratory-confirmed SARS-CoV-2 infection; SARS-CoV-2 infection within 4 weeks prior to screening; and/or history of severe course of COVID-19
* If female, pregnancy (defined as positive beta-HCG blood test and/or positive urine pregnancy test), breast-feeding

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Treatment part I: Photosensitivity Index (PI) at 10 minutes post UV irradiation under Condition 1 | On-drug Day 8
  The PI is calculated as the ratio of the minimal erythema dose (MEDbaseline) measured on Day -2 at 10 minutes post-irradiation to the corresponding MEDon-drug measured on Day 8 at 10 minutes post-irradiation.
  Condition 1 is Full range solar ultraviolet B/ultraviolet A (UVB/UVA) [290 to 400 nm] exposure.
Treatment part I: Photosensitivity Index (PI) at 1 hour post UV irradiation under Condition 1 | On-drug Day 8
  The PI is calculated as the ratio of the minimal erythema dose (MEDbaseline) measured on Day -2 at 1 hour post-irradiation to the corresponding MEDon-drug measured on Day 8 at 1 hour post-irradiation.
  Condition 1 is full range solar UVB/UVA [290 to 400 nm] exposure.
Treatment part I: Photosensitivity Index (PI) at 24 hours post UV irradiation under Condition 1 | On-drug Day 9
  The PI is calculated as the ratio of the minimal erythema dose (MEDbaseline) measured on Day -1 at 24 hours post-irradiation to the corresponding MEDon-drug measured on Day 9 at 24 hours post-irradiation.
  Condition 1 is a Full range solar UVB/UVA [290 to 400 nm] exposure.
Treatment part I: Photosensitivity Index (PI) at 10 minutes post UV irradiation under Condition 2 | On-drug Day 8
  The PI is calculated as the ratio of the minimal erythema dose (MEDbaseline) measured on Day -2 at 10 minutes post-irradiation to the corresponding MEDon-drug measured on Day 8 at 10 minutes post-irradiation.
  Condition 2 is a UVA only [320 to 400 nm] exposure.
Treatment part I: Photosensitivity Index (PI) at 1 hour post UV irradiation under Condition 2 | On-drug Day 8
  The PI is calculated as the ratio of the minimal erythema dose (MEDbaseline) measured on Day -2 at 1 hour post-irradiation to the corresponding MEDon-drug measured on Day 8 at 1 hour post-irradiation.
  Condition 2 is a UVA only [320 to 400 nm] exposure.
Treatment part I: Photosensitivity Index (PI) at 24 hours post UV irradiation under Condition 2 | On-drug Day 9
  The PI is calculated as the ratio of the minimal erythema dose (MEDbaseline) measured on Day -1 at 24 hours post-irradiation to the corresponding MEDon-drug measured on Day 9 at 24 hours post-irradiation.
  Condition 2 is a UVA only [320 to 400 nm] exposure.

SECONDARY OUTCOMES:
Treatment part I & part II: Minimum Erythema Dose (MED) percent change from baseline at 10 minutes, 1 hour, and 24 hours postirradiation measured under Condition 1 and Condition 2 | Baseline (Day -2 to Day -1) and on-drug (Day 8 to Day 9)
  Condition 1 is full range solar UVB/UVA [290 to 400 nm] exposure and condition 2 is a UVA only [320 to 400 nm] exposure.
Treatment part I & part II: Evaluation of local skin reactions following exposure to UV irradiation at 10 minutes, 1 hour, 24 hours, 48 hours, and 72 hours postirradiation under Condition 1, Condition 2, and Condition 3 | At Baseline (Day -2 to Day 1 pre-dose) and on-drug (Day 8 to Day 11)
  Condition 1 is full range solar UVB/UVA [290 to 400 nm] exposure, condition 2 is a UVA only [320 to 400 nm] exposure and condition 3 is a full solar range UVB/UVA + UVA [16 J/cm2] exposure.
Treatment part I: Assessment of Plasma pharmacokinetic parameter of SAR441566: Cmax | Day 8 to Day 11
  Maximum plasma concentration observed
Treatment part I: Assessment of Plasma pharmacokinetic parameter of SAR441566: Tmax, | Day 8 to Day 11
  Time to reach Cmax
Treatment part I: Assessment of Plasma pharmacokinetic parameter of SAR441566: AUC0-tau | Day 8 to Day 9
  Area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (0 to 24 hours)
Treatment part I: Number of participants with adverse events (AE) and treatment-emergent adverse events (TEAEs) | Up to Day 20
  Assessment of adverse events (AE) / treatment-emergent adverse events (TEAE) including serious adverse event (SAE) and adverse event of special interests (AESI)
Treatment part II: Photosensitivity Index (PI) at 10 minutes post UV irradiation under Condition 1 | On-drug Day 8
  Condition 1 is full range solar UVB/UVA [290 to 400 nm] exposure.
Treatment part II: Photosensitivity Index (PI) at 1 hour post UV irradiation under Condition 1 | On-drug Day 8
  Condition 1 is full range solar UVB/UVA [290 to 400 nm] exposure.
Treatment part II: Photosensitivity Index (PI) at 24 hours post UV irradiation under Condition 1 | On-drug Day 9
  Condition 1 is full range solar UVB/UVA [290 to 400 nm] exposure.
Treatment part II: Photosensitivity Index (PI) at 10 minutes Condition 2 | On-drug Day 8
  Condition 2 is a UVA only [320 to 400 nm] exposure.
Treatment part II: Photosensitivity Index (PI) at 1 hour post UV irradiation under Condition 2 | On-drug Day 8
  Condition 2 is a UVA only [320 to 400 nm] exposure.
Treatment part II: Photosensitivity Index (PI) at 24 hours post UV irradiation under Condition 2 | On-drug Day 9
  Condition 2 is a UVA only [320 to 400 nm] exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- TKL Research, Inc. Site Number : 8400001, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PDY16917 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25320&tenant=MT_SNY_9011